CLINICAL TRIAL: NCT00222495
Title: A Comparative Study of New Medications for Psychosis in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: AstraZeneca (Industry); Jensen, Jonathan B., M.D. (Individual)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0205M26041
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Psychotic Disorders; Schizophrenia; Schizophreniform Disorders; Schizoaffective Disorders
Keywords: Psychotic Disorders in adolescents; Schizophrenia in adolescents; Schizophreniform Disorders in adolescents; Schizoaffective Disorders in adolescents
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Quetiapine Fumarate; Olanzapine; Risperidone

INTERVENTIONS:
Drug: quetiapine
Drug: olanzapine
Drug: risperidone

SUMMARY:
The overall goal of this study is to determine the efficacy and tolerability of three atypical antipsychotic medications (risperidone, olanzapine, and quetiapine) in the treatment of adolescents with psychosis. It is hypothesized that the three medications will be equally effective in reducing the symptoms of psychosis.

DETAILED DESCRIPTION:
The purpose of this study is to compare the efficacy and tolerance of three atypical antipsychotics, which are medications that have been in use for about the last 10 years, in the treatment of psychosis in adolescents. Efficacy refers to how well the medications work in decreasing symptoms associated with schizophrenia, and tolerance refers to the level of side effects and the compliance with taking the medications. All three medications have demonstrated efficacy in treating psychosis without causing extra pyramidal side effects (uncontrolled muscle movements) that are associated with typical, or older antipsychotic medications. Young people may be at a greater risk for side effects from the typical antipsychotic medications. There are studies of the efficacy and tolerance among patients under 18-years-old taking the three drugs in this study: risperidone, olanzapine, and quetiapine. However, at this time there is little data available comparing these three medications. This study is an open-label, random assignment, 12-week study to assess the efficacy and tolerance of these three atypical antipsychotic medications in the treatment of adolescents (ages 12-18) with schizophrenia or psychosis. The participants will be informed of which medication she/he is taking, and will be assigned to the medication randomly (based on chance rather than choice).

There are additional theoretical beliefs in regard to this study as well. A secondary hypothesis of this study is that quetiapine will have less extra pyramidal side effects (EPS) and less prolactin-related side effects than risperidone. A third hypothesis is that quetiapine will lead to less weight gain than olanzapine and risperidone. Finally, it is hypothesized that because of the fewer side effects, quetiapine will be better tolerated than risperidone and olanzapine.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are between the ages of 12-18 and have a diagnosis of a psychotic illness.
2. Subject currently meets criteria for one of the following disorders: schizophrenia, schizoaffective disorder (mainly schizophrenic), schizophreniform disorder, and psychosis NOS.
3. Subject is in good physical health and not suffering from any medical disorder that might mimic psychosis or lead to medical difficulty with the study medications.
4. If subject is taking antipsychotic medication before study entry, their medicine will be discontinued for 1-4 days depending on symptoms.

Exclusion Criteria:

1. Subject has a medical disorders that would interfere with the study, such as epilepsy, thyroid disease, liver disease, AIDS, etc.
2. Subject currently has substance dependence.
3. Subject is talking a medication that inhibits or induces the cytochrome P450 3A4 (specific medications listed in Appendix of protocol).

3. Subject meets criteria for brief psychosis or mood disorder with psychotic features.

4. Female subject is pregnant or nursing.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30
Dates: Start 2002-08; Study Completion 2006-08

PRIMARY OUTCOMES:
SCI-PANSS = Structured Clinical Interview - Positive and Negative Syndrome Scale
CGI = Clinical Global Impressions
GAF = Global Assessment of Functioning Scale

SECONDARY OUTCOMES:
Neuropsychological assessment battery
Calgary Depression Symptoms for Schizophrenia
AIMS = Abnormal Involuntary Movement Scale
Barnes-Akathisia Rating Scale
SAS = Simpson Angus Scale

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Jensen, M.D., Principal Investigator — University of Minnesota; S. Charles Schulz, M.D., Study Director — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States